CLINICAL TRIAL: NCT06551220
Title: HER2 Heterogeneity and Its Impact on Benefit from Trastuzumab Deruxtecan in Metastatic Breast Cancer
Brief Title: Efficacy of Trastuzumab Deruxtecan in Metastatic Breast Cancer with Different HER2 Expression Patterns
Acronym: HEROIC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yutian Zou, Assistant Professor, Sun Yat-sen University
Other Study IDs: SYSUCC-B2022-617-X01
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; Trastuzumab Deruxtecan; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin section
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trastuzumab Deruxtecan
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — The patients received Trastuzumab Deruxtecan at a dose of 5.4 mg/kg every 3 weeks until disease progression or unacceptable adverse effects occurred.

SUMMARY:
The purpose of this observational study is to learn about the HER2 heterogeneity and its impact on benefit from trastuzumab deruxtecan in metastatic breast cancer. The main question it aims to answer is:

- Does the heterogeneity of HER2 expression level and spatial distribution in different tissues affect the efficacy of trastuzumab deruxtecan in metastatic breast cancer?

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or locally unresectable breast cancer;
* Treated with T-DXd (DS-8201, trastuzumab deruxtecan) regardless of line of therapy, HR, and HER2 expression level;
* HER2 immunohistochemistry staining information of the primary lesion or metastatic/recurrent lesion;
* Measurable lesions with treatment response results that can be evaluated through imaging examinations;
* Able to follow up with the latest progression-free survival or overall survival.

Exclusion Criteria:

* Patients with missing basic clinical information or HER2 immunohistochemistry staining information;
* Patients with missing pathological results for both primary and metastatic/recurrent lesions;
* Patients with no measurable lesions and unable to evaluate T-DXd treatment response;
* Discontinue T-DXd therapy for unacceptable adverse events or other reasons;
* Patients lost to follow-up after T-DXd treatment.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multicenter, retrospective study led by the Sun Yat-sen University Cancer Center. A total of 16 centers are planned to participate in the study, and it aims to include patients with advanced or locally unresectable breast cancer who have received treatment with T-DXd.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of T-DXd treatment initiation until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 60 months.
  Progression-free survival (PFS) is defined as the time from T-DXd treatment initiation to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of T-DXd treatment initiation until the date of death from any cause, assessed up to 60 months.
  Overall survival (OS) is defined as the time from treatment initiation to death from any cause.

OTHER OUTCOMES:
Objective response rate (ORR) | From screening and every 2-6 weeks up to progressive disease, or unacceptable toxicity, assessed up to 60 months.
  The Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) was used as the standard for evaluating treatment response to T-DXd. The response was evaluated based on the change in the tumor relative to baseline and was categorized as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). Objective response rate (ORR) is defined as the proportion of patients who achieved CR or PR.
Disease control rate (DCR) | From screening and every 2-6 weeks up to progressive disease, or unacceptable toxicity, assessed up to 60 months.
  The Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) was used as the standard for evaluating treatment response to T-DXd. The response was evaluated based on the change in the tumor relative to baseline and was categorized as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). Disease control rate (DCR) was defined as the proportion of patients who achieved CR, PR, or SD.
Clinical benefit rate (CBR) | From screening and every 2-6 weeks up to progressive disease, or unacceptable toxicity, assessed up to 60 months.
  The Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) was used as the standard for evaluating treatment response to T-DXd. The response was evaluated based on the change in the tumor relative to baseline and was categorized as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). The clinical benefit rate (CBR) was defined as the proportion of patients who achieved CR, PR, or SD for at least 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Xie, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (23):
- China (21):
  - Fujian Cancer Hospital, Fujian Medical University, Fuzhou, Fujian
  - The 10th Affiliated Hospital of Southern Medical University, Dongguan, Guangdong
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The Sixth Affiliated Hospital, School of Medicine, South China University of Technology., Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Yuebei People's Hospital of Shantou University, Shaoguan, Guangdong
  - National Cancer Center Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Changde Hospital, Xiangya School of Medicine, Central South University, Changde, Hunan
  - Hunan Cancer Hospital/The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital, Hengyang Medical School, University of South China, Hengyang, Hunan
  - Affiliated Cancer Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Xinhua Hospital Afliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Country not given (2):
  - Cancer Hospital of Shantou University Medical College
  - The Affiliated Panyu Central Hospital, Guangzhou Medical University